CLINICAL TRIAL: NCT05450705
Title: A Phase 3 Open-Label Immunogenicity and Safety Study of 2-Dose Regimens of a 9vHPV Vaccine (V503) in Chinese Girls 9 Through 14 Years of Age With a Comparison to 3-Dose Regimen of V503 in Chinese Women 20 Through 26 Years of Age
Brief Title: V503 in Chinese Girls 9-14 Years Old Versus Chinese Women 20-26 Years Old (V503-071)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-071; V503-071 (Other: Merck)
Record Dates: First submitted 2022-06-28; First posted 2022-07-11 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 9 to 14 Years Old: Day 1 and Month 6 (Experimental): Chinese females 9 to 14 years old will receive a 0.5 mL intramuscular (IM) injection of 9-valent HPV (9vHPV) vaccine on Day 1 and Month 6
  Interventions: Biological: 9vHPV vaccine
- 9 to 14 Years Old: Day 1 and Month 12 (Experimental): Chinese females 9 to 14 years old will receive a 0.5 mL iIM injection of 9-valent HPV (9vHPV) vaccine on Day 1 and Month 12
  Interventions: Biological: 9vHPV vaccine
- 20 to 26 Years Old: Day 1, Month 2 and Month 6 (Experimental): Chinese females 20 to 26 years old will receive a 0.5 mL IM injection of 9-valent HPV (9vHPV) vaccine on Day 1, Month 2 and Month 6
  Interventions: Biological: 9vHPV vaccine

INTERVENTIONS:
Biological: 9vHPV vaccine — A 9-valent HPV vaccine (Types 6, 11, 16, 18, 31, 33, 45, 52, and 58) will be administered as a 0.5 mL IM injection.
  Other Names: V503; GARDASIL9™

SUMMARY:
This study aims to demonstrate that a 2-dose regimen of the 9-Valent Human Papillomavirus (9vHPV) vaccine (GARDASIL™9, V503) induces non-inferior competitive Luminex immunoassay (cLIA) geometric mean titers (GMTs) to each of the 9vHPV vaccine types in Chinese girls 9 through 14 years of age compared to a 3-dose regimen in Chinese women 20 through 26 years of age. The primary hypothesis is that a 2-dose regimen has a non-inferiority margin of 0.67 in the GMT ratio (girls vs. women) for each HPV type.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Is a healthy Chinese female.
* Is not a woman of childbearing potential (WOCBP); or is a WOCBP who has not had sex with males or has had sex with males and used effective contraception during Day 1 through 1 month post last dose.

Exclusion Criteria:

* Has a history of known prior vaccination with an HPV vaccine.
* Has a history of severe allergic reaction that required medical intervention.
* Has a known thrombocytopenia or coagulation disorder that would contraindicate IM injections.
* Has a history of abnormal Pap test or external genital wart, vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, anal intraepithelial neoplasia, vulvar cancer, vaginal cancer, or anal cancer.
* Has a history of a positive test for HPV.
* Has received immune globulin or blood-derived products in the past 6 months or plans to receive any before one month post last dose.
* Has a history of splenectomy, is currently immunocompromised, or has been diagnosed with immunodeficiency, human immunodeficiency virus, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition.
* Has received immunosuppressive therapy in the past year, excluding inhaled, nasal, or topical corticosteroids and certain regimens of systemic corticosteroids.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1500 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2029-08-03 (Estimated); Study Completion 2029-08-03 (Estimated)

PRIMARY OUTCOMES:
Stage I: Competitive Luminex immunoassay (cLIA) Geometric Mean Titers (GMTs) to 9 vaccine types of 9vHPV vaccine | One month after last dose (Up to Month 13)
  cLIA GMT to each of 9 vaccine types of 9vHPV vaccine. The GMT for each HPV type will be reported in mMU/mL.
Stage II: cLIA GMTs to 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age | Up to Month 84
  cLIA GMT to each of 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age. The GMT for each HPV type will be reported in mMU/mL.
Stage II: cLIA seropositivity percentages to 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age | Up to Month 84
  cLIA seropositivity to each of 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age. The percentage of participants who are seropositive for each HPV type will be summarized.

SECONDARY OUTCOMES:
Stage I: cLIA seroconversion percentages to 9 vaccine types of 9vHPV vaccine | One month after last dose (Up to Month 13)
  cLIA seroconversion to each of 9 vaccine types of 9vHPV vaccine. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage I: Immunoglobulin G Luminex immunoassay (IgG LIA) GMTs to 9 vaccine types of 9vHPV vaccine at one month post last dose | One month after last dose (Up to Month 13)
  IgG LIA GMT to each of 9 vaccine types of 9vHPV vaccine at one month post last dose. The GMT for each HPV type will be reported in mMU/mL.
Stage I: IgG LIA seroconversion percentages to 9 vaccine types of 9vHPV vaccine | One month after last dose (Up to Month 13)
  IgG LIA seroconversion to each of 9 vaccine types of 9vHPV vaccine. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage I: Percentage of participants experiencing solicited injection-site adverse events (AEs) | Day 1 through Day 8 following any study vaccination
  An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Solicited injection-site AEs such as erythema, swelling, pain, and induration at the injection site will be recorded.
Stage I: Percentage of participants experiencing solicited systemic AEs | Day 1 through Day 8 following any study vaccination
  An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Systemic AEs are those not categorized as injection-site AEs.
Stage I: Percentage of participants experiencing serious AEs (SAEs) Up to Month 13 | Up to Month 13
  A SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.
Stage II: Percentage of participants experiencing SAEs Up to Month 84 | Month 18 up to Month 84
  A SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.
Stage II: IgG LIA GMTs to 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age | Up to Month 84
  IgG LIA GMT to each of 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age. The GMT for each HPV type will be reported in mMU/mL.
Stage II: IgG LIA seropositivity percentages to 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age | Up to Month 84
  IgG LIA seropositivity to each of 9 vaccine types of 9vHPV vaccine in girls 9 through 14 years of age. The percentage of participants who are seropositive for each HPV type will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- China (2):
  - Jiangshan Center for Disease Control and Prevention ( Site 0001), Quzhou, Zhejiang
  - Yuhuan Center for Disease Control and Prevention ( Site 0002), Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php